CLINICAL TRIAL: NCT07038031
Title: Nutrition in Action: Service-Learning Project
Acronym: NA_SL
Status: Not yet recruiting | Type: Observational
Sponsor: University of Vic - Central University of Catalonia (Other)
Collaborators: Fundació sant tomàs (Unknown); Creu Roja Osona (Unknown); Centre Formació Persones Adultes Montseny (Unknown); Centre Formació Persones Adultes Miquel Martí i Pol (Unknown); Adults Training Centers (Unknown)
Responsible Party: Sponsor
Other Study IDs: Nutrition_SLp_UVic-UCC
Record Dates: First submitted 2025-05-28; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Skills Acquisition; Satisfaction
Keywords: Service-learning; Skills; Food habits; Higher education
MeSH Terms: conditions — Personal Satisfaction; Feeding Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention group: The intervention group are university students from the food education strategies (FES) subject from the 6th term of the Human Nutrition and Dietetics Degree (ND) of the Faculty of Health and Welfare Sciences (FCSB) of the University of Vic-Central University of Catalonia (UVic-UCC).
  They develop the service learning project to promote a healthy food habits in diferent social organitzations of the territory. It consists to do an interview to identify nutritional educational needs, and do 3 nutritional workshops to participants from this organitzations. Each workshop has 1 hour, and is addreced to a small group of participants (8-15 maximum), always with the supervision of the professional of the social organitzation.
  Interventions: Behavioral: Promotion a food habits

INTERVENTIONS:
Behavioral: Promotion a food habits — They develop the service learning project to promote a healthy food habits in diferent social organitzations of the territory. It consists to do an interview to identify nutritional educational needs, and do 3 nutritional workshops to participants from this organitzations. Each workshop has 1 hour, and is addreced to a small group of participants (8-15 maximum), always with the supervision of the professional of the social organitzation.

SUMMARY:
Service-learning methodology (SL) combines training and community processes in a single project where participants are trained while working on real needs of the environment with the aim of improving it. This methodology enhances the professional skills of the students, their personal and competence development, and develops a deeper sense of civic responsibility.

The Human Nutrition and Dietetics Degree (ND) of the Faculty of Health and Welfare Sciences (FCSB) of the University of Vic-Central University of Catalonia decided to incorporate this methodology, according to University's training model, with the aim of generating learning situations that allow them to act, reflect and solve problems based on significant learning. We applied SL in the subject of Food Education Strategies designing and implementing a small food education program with 1 contact to detect the needs of the users, and 3 educational sessions. The implementation of the SL is based on the SL guide proposed by the Service Learning Network of Catalan Universities and we make it with 4 local social entities.

The teacher responsible for the SL is coordinated with responsibles from entities who act as facilitators, authorizing the collection of data from the people of the entities, recruiting, informing and collecting the willingness to participate from the users.

We plan to study the experience of participating in the SL activity in terms of student acquisition of skills and satisfaction of all the parties involved, based on an observational study carried out during 4 academic years (2025-2029).

Through convenience sampling, a participation of 65 people is expected (20 students, 40 users, 5 responsible from entities).

Data collection plans to compile information on: a.Experience of the SL of the university student body. b. Assessments of the users and responsibles from entities on the impact, quality and satisfaction with the SL activity. c. Proposal for improving the SL activity with the entities using the rubric for self-assessment and improvement of SL projects.

Data collection will take place at the end of the activity using the REDCap platform (Research Electronic Data Capture) and the statistic analysis is planned using the SPSS statistical program.

DETAILED DESCRIPTION:
The local social entities are: the St. Tomàs Foundation, the Vic Red Cross, the Miquel Martí i Pol Adult Education Center and the Montseny Adult Education Center.

The students developed content and resources to adapt the dietary advice to one of the 4 entities in small groups of 3-5 people. They prepared the material during the subject guided by the teacher taking into account the characteristics of the users (elderly people living alone, people with disabilities, multicultural diversity).

The entities welcome the university students and the managers of each entity guide them in developing the sessions. At the end of the Vic Classroom activity, the entities evaluate the students and the activity.

ELIGIBILITY:
Inclusion Criteria:

* University students enrolled in the Food Education Strategies subject of the Nutrition and Dietetics Degree at the UVic-UCC.

Exclusion Criteria:

* Online students.
* Students who do not voluntarily agree to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All students enrolled in the Food Education Strategies subject, who are doing the Nutrition and Dietetics Degree in a presencial modality, in the UVic-UCC.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Service-Learning methodology | Through study completion, an average of 1 month
  We want to describe: Attitudes toward self, attitudes toward school and learning, civic engagement, social skills, and academic performance, using a validated questionnaire for an spanish university' students from León-Carrascosa, Sánchez-Serrano, i Belando-Montoro (2020). It is validated in the Spanish university population and includes a total of 35 items to which students must respond on a 1 to 5 Likert-type scale (1 indicates not at all, and 5 indicates completely).

SECONDARY OUTCOMES:
Satisfaction with Service-learning | Through study completion, an average of 1 month
  We would like to ask to the participants their satisfaction with the activity. We use a Visual Analog Scale we 0 is very bad experience, and 10 is very good experience.

CONTACTS AND LOCATIONS:
Locations (1):
- UVic-UCC, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The rubric is a tool designed to facilitate self-evaluation and improvement of service-learning experiences. Twelve dynamics are presented, organized into three sections-basic, pedagogical, and organizational-and four levels for each of the dynamics. — https://aprenentatgeservei.cat/wp-content/uploads/guies/aps_autoevaluacio_cat_mini_IMPA4.pdf